CLINICAL TRIAL: NCT06485986
Title: Frontosubthalamic Network Dynamics and Their Modulation During Impulse Control and Decision Making in Parkinson's Disease
Brief Title: Frontosubthalamic Networks in Parkinson's Disease.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: PID14888
Record Dates: First submitted 2024-06-26; First posted 2024-07-03 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Parkinson Disease; Impulse Control Disorder
Keywords: Deep brain stimulation
MeSH Terms: conditions — Parkinson Disease; Disruptive, Impulse Control, and Conduct Disorders

STUDY DESIGN:
Intervention Model Description: Two groups of patients will be recruited:
  * Parkinson's disease patients treated with deep brain stimulation and no impulse control disorder
  * Parkinson's disease patients treated with deep brain stimulation and impulse control disorder (an increase in QUIP-RS after surgery)
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parkinson's Disease DBS, no Impulse Control Disorder (Active Comparator): Patients with Parkinson's disease who are treated with deep brain stimulation (DBS) but have not developed impulsive or compulsive behaviours will undertake a computerised task with their DBS turned on and off with simultaneous magnetoencephalography. After each experiment, normal therapy will be resumed.
  Interventions: Other: DBS on/off
- Parkinson's Disease DBS, with Impulse Control Disorder (Experimental): Patients with Parkinson's disease who are treated with deep brain stimulation (DBS) who have developed impulsive or compulsive behaviours will undertake a computerised task with their DBS turned on and off with simultaneous magnetoencephalography. After each experiment, normal therapy will be resumed.
  Interventions: Other: DBS on/off

INTERVENTIONS:
Other: DBS on/off — DBS will be turned on and off for experimental periods to compare the effect of DBS on behaviour.

SUMMARY:
The goal of this experimental study with is to understand the underlying mechanisms behind the increase in impulsivity seen in some patients that undergo deep brain stimulation of the subthalamic nucleus for Parkinson's Disease. The main questions it aims to answer are:

What are the distributed network effects of deep brain stimulation to the subthalamic nucleus? How does this correlate with increased impulsivity? Can alternative stimulation settings be used to minimize these?

Participants will complete decision-making tasks whilst their deep brain stimulation devices are turned on and off with simultaneous magnetoencephalography recordings (a type of non-invasive brain scan that measures brain activity in real-time)

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 18 years or above.
* Diagnosed with Parkinson's disease who have required implanted STN electrodes for DBS in addition to their dopamine replacement therapy.
* Diagnosed with or without (control group) impulse control disorders since the diagnosis of Parkinson's Disease.
* Participant willing and able to sit in the MEG scanner and follow instructions.
* Participant willing and able to delay their morning dose of dopamine replacement therapy for up to four hours (180 minutes experimental time + journey time).

Exclusion Criteria:

* Patients with extreme language barrier that cannot understand the purpose or instructions of the study despite the use of an interpreter.
* Other implanted medical devices that may cause artefacts during MEG recordings.
* Participants with a history of co-morbid neurological disorders.
* Participant enrolled onto another clinical trial related to a neurological disorder (including Parkinson's disease) that may interfere with the results of this study.
* Participants who are unable to sit still in a MEG scanner for the duration of this experiment e.g. patients with chronic pain or osteoarthritis. This will be assessed with their primary clinician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Identify effect of therapeutic STN-DBS on frontosubthalamic networks in PD related ICDs during decision making and impulse control | 12 months
  Correlation between response time and accuracy with electrophysiological signatures of neural activity.

CONTACTS AND LOCATIONS:
Locations (1):
- John Radcliffe Hospital, Oxford, United Kingdom

REFERENCES:
- [Background] Herz DM, Frank MJ, Tan H, Groppa S. Subthalamic control of impulsive actions: insights from deep brain stimulation in Parkinson's disease. Brain. 2024 Nov 4;147(11):3651-3664. doi: 10.1093/brain/awae184. PMID 38869168
- [Background] Eraifej J, Cabral J, Fernandes HM, Kahan J, He S, Mancini L, Thornton J, White M, Yousry T, Zrinzo L, Akram H, Limousin P, Foltynie T, Aziz TZ, Deco G, Kringelbach M, Green AL. Modulation of limbic resting-state networks by subthalamic nucleus deep brain stimulation. Netw Neurosci. 2023 Jun 30;7(2):478-495. doi: 10.1162/netn_a_00297. eCollection 2023. PMID 37397890